CLINICAL TRIAL: NCT04174573
Title: Efficacy of Group Therapy With Transcranial Direct Current Stimulation on Balance and Quality of Life in Patients With Parkinson's Disease: A Single Blind, Multi-centre, Randomized Clinical Study
Brief Title: Group Therapy With Transcranial Direct Current Stimulation in Patients With Parkinson's Disease
Acronym: GTBQ-PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1240-0949
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
Keywords: tDCS; Quality of Life; Parkinson Disease; Neuronal Plasticity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group therapy only (GTO) (Experimental): Patients in GTO group will receive structured group therapy programme
  Interventions: Other: GTO
- Group therapy with tDCS (GT-tDCS) (Experimental): Patients in this group will receive group therapy along-with tDCS intervention
  Interventions: Other: GT-tDCS

INTERVENTIONS:
Other: GTO — 1. Forward direction activity: Balance activity in forward direction on wooden balance board (5 reps X 3 sets X 2 days in a week, for 6 weeks)
  2. Backward direction activity: Balance activity in backward direction on wooden balance board (5 reps X 3 sets X 2 days in a week, for 6 weeks)
  3. Sideways direction activity: Balance activity in sideways direction on wooden balance board (5 reps X 3 sets X 2 days in a week, for 6 weeks)
  Arms: Group therapy only (GTO)
Other: GT-tDCS — 1. Group therapy
     1. Forward direction activity: Balance activity in forward direction on wooden balance board (5 reps X 3 sets X 2 days in a week, for 6 weeks)
     2. Backward direction activity: Balance activity in backward direction on wooden balance board (5 reps X 3 sets X 2 days in a week, for 6 weeks)
     3. Sideways direction activity: Balance activity in sideways direction on wooden balance board (5 reps X 3 sets X 2 days in a week, for 6 weeks)
  2. tDCS Left anodal and right cathodal tDCS : Anode- F3, Cathode- Right Supra orbital area, Intensity- 2mA, Duration- 30 minutes, once in a week for 6 weeks
  Arms: Group therapy with tDCS (GT-tDCS)

SUMMARY:
To determine the effectiveness of group therapy along with transcranial direct current (tDCS) stimulation on motor symptoms, balance and quality of life in patients with Parkinson's disease(PD). 128 patient with PD will be recruited by the cluster sampling method for the two group pretest-posttest randomized controlled trial. The patient with PD will be allocated in two groups, Group therapy only (GTO) group and Group therapy with tDCS (GT-tDCS) treatment group by block randomization technique. Both GTO group and GT-tDCS group will receive the structured group therapy programme for one hour duration, twice a week for 6-weeks. In addition to the structured group therapy programme, GT-tDCS group will receive 20 minutes of tDCS application once a week for the 6-week duration. Data will be analysed at baseline, 3 weeks and 6 weeks of post intervention.

DETAILED DESCRIPTION:
Introduction:

Parkinson disease (PD) occurs due to degenerative changes in the nervous system, dysfunctions of basal ganglia. Patients affected with PD survive with the postural and mobility impairments that leads to impaired quality of life. Medical and surgical procedures do not provide the patient with a fully effective response.1 Literature suggests that physical therapy can improve the quality of life and balance function in patients with PD. Group therapy (GT) intervention is found to be significant intervention in aspects of mobility in various neurological conditions. GT have been used as part of supervised group rehabilitation to improve balance in patient with PD.2 Patients with PD have difficulties with learning of new motor skills, but recent neuro-modulatory techniques by noninvasive brain stimulation helps to facilitate motor skills and regulate neuroplasticity.

Transcranial direct current stimulation (tDCS) is a therapeutic device that is used to improve motor symptoms of PD, when applied to primary motor cortex M1. Anodal tDCS can increase M1 excitability, reduce cortical inhibition and results in improved functional performance. When combined with other exercise training, it provides longer lasting effect in motor function.3 However, no studies have investigated the concurrent use of anodal tDCS and group therapy intervention in patient with PD.

The aims of this study are to determine the effects of a 3 weeks concurrent GT and anodal tDCS intervention on measures of static and dynamic balance and to evaluate any long-term effects.

The investigators hypothesize that the combination of group therapy and anodal tDCS will improve balance and quality of life than group therapy or anodal tDCS alone.

Methodology of the proposed study Ethical statement and Subject recruitment The study protocol was approved by the institutional research advisory committee (RAC) and registered under the Universal Trial Number (UTN), U1111-1240-0949. The protocol will be registered under ClinicalTrials.gov, under World Health Organization International Clinical Trials Registry Platform and then the study will be submitted for the ethical approval by institutional ethics committee of Maharishi Markandeshwar Deemed to Be University, Mullana, and Haryana with unique reference number. The study will be executed in accordance with the principles of the Declaration of Helsinki (Revised, 2013) and National ethical guidelines for Biomedical and Health research involving human participants by Indian council for medical research (ICMR, 2017). The purpose of the study will be clearly explained to the patient with PD. Written informed consent form will be obtained from the recruited patients. The study will be performed between October, 2019 and March, 2022.

Inclusion Criteria

* Presence of mild neurocognitive disorders was based on the validated Montreal Cognitive Assessment (MoCA) cutoff scores (<23.5)
* Based on the Hoehn-Yahr Stage (HYS) staging, severity of PD was categorized as mild (HYS 1&2), moderate (HYS 3) and severe (HYS 4&5). Patient with PD with mild and moderate will be recruited Exclusion Criteria
* Patient with PD with associated comorbidities such as stroke, uncontrolled diabetes, sensory impairments such as hearing, vision, etc.
* Patient with PD who is not willing to participate in the study Total of X patient with PD will be screened and through convenience sampling method, 34 children will be selected based on the inclusion criteria for the two group pretest-posttest randomized controlled trial. Demographic data will be recorded for all the recruited patient with PD. The patient with PD will be allocated in two groups, Group therapy only (GTO) group and Group therapy with tDCS (GT-tDCS) treatment group by block randomization technique. The total required sample size of, n=128 will be randomized into both the groups. According to it, there will be four blocks, with the matrix design of 4 × 32, where32 being rows. Each row could have four blocks, with one chit (SNOSE - sequentially numbered, opaque sealed, envelopes) in each block containing either the name of GTO group or GT-tDCS group. Total four chits (2 chits for each group) will be assigned to each row and then patient with PD will be allotted to one of the two group based on the randomly chosen chit (SNOSE). Once the entire first row will be allotted, then the next row block will be opened for enrolment. The advantage of this method of randomization is that the number of patients assigned to each group over time would have been approximately equal. By this the unequal allocation of sample size, will be avoided. The concealed allocation of patient with PD to the treatment groups will be explained by using SNOSE.

Both GTO group and GT-tDCS group will receive the structured group therapy programme for one hour duration, twice a week for 6-weeks. In addition to the structured group therapy programme, GT-tDCS group will receive 20 minutes of tDCS application once a week for the 6-week duration. Outcomes will be used to analysed the data at baseline, 3 weeks and 6 weeks post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Presence of mild neurocognitive disorders was based on the validated Montreal Cognitive Assessment (MoCA) cutoff scores (<23.5)
* Based on the Hoehn-Yahr Stage (HYS) staging, severity of PD was categorized as mild (HYS 1&2), moderate (HYS 3) and severe (HYS 4&5). Patient with PD with mild and moderate will be recruited

Exclusion Criteria:

* Patient with PD with associated comorbidities such as stroke, uncontrolled diabetes, sensory impairments such as hearing, vision, etc.
* Patient with PD who is not willing to participate in the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-06-06 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Movement Disorders Society Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS). | Change will be measured at baseline, 3 weeks and after 6 weeks of intervention
  The Unified Parkinson Disease Rating Scale, designed to monitor the burden and extent of Parkinson's disease. o-4 score, lower the score indicates normal, higher the scores indicate greater impact of PD symptoms.
Parkinson's Disease Questionnaire with 39 items | Change will be measured at baseline, 3 weeks and after 6 weeks of intervention
  The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month.
  Assesses how often patients experience difficulties across the 8 quality of life dimensions.
  Assesses impact of Parkinson's Disease (PD) on specific dimensions of functioning and well-being. Each dimension total score ranges from 0 (never have difficulty) to 100 (always have difficulty). lower score reflect better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Adarsh K Srivastav, MPT, Principal Investigator — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] King LA, Wilhelm J, Chen Y, Blehm R, Nutt J, Chen Z, Serdar A, Horak FB. Effects of Group, Individual, and Home Exercise in Persons With Parkinson Disease: A Randomized Clinical Trial. J Neurol Phys Ther. 2015 Oct;39(4):204-12. doi: 10.1097/NPT.0000000000000101. PMID 26308937
- [Result] Lattari E, Costa SS, Campos C, de Oliveira AJ, Machado S, Maranhao Neto GA. Can transcranial direct current stimulation on the dorsolateral prefrontal cortex improves balance and functional mobility in Parkinson's disease? Neurosci Lett. 2017 Jan 1;636:165-169. doi: 10.1016/j.neulet.2016.11.019. Epub 2016 Nov 9. PMID 27838447
- [Result] Renner CIe, Outermans J, Ludwig R, Brendel C, Kwakkel G, Hummelsheim H. Group therapy task training versus individual task training during inpatient stroke rehabilitation: a randomised controlled trial. Clin Rehabil. 2016 Jul;30(7):637-48. doi: 10.1177/0269215515600206. Epub 2015 Aug 27. PMID 26316552
- [Result] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for idiopathic Parkinson's disease. Cochrane Database Syst Rev. 2016 Jul 18;7(7):CD010916. doi: 10.1002/14651858.CD010916.pub2. PMID 27425786
- [Result] Nero H, Franzen E, Stahle A, Benka Wallen M, Hagstromer M. Long-Term Effects of Balance Training on Habitual Physical Activity in Older Adults with Parkinson's Disease. Parkinsons Dis. 2019 Aug 7;2019:8769141. doi: 10.1155/2019/8769141. eCollection 2019. PMID 31485305